CLINICAL TRIAL: NCT00004367
Title: Vestibular Dysfunction In Adult Patients With Panic Disorder With or Without Agoraphobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pittsburgh (Other)
Purpose: Diagnostic
Other Study IDs: 199/11945; UPITTS-9504279605
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Anxiety Disorder; Panic Disorder
Keywords: anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; panic disorder; rare disease
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Procedure: Clinical vestibular tests

SUMMARY:
OBJECTIVES: I. Determine whether the prevalence of abnormalities on clinical vestibular (balance) tests is higher in panic disorder with agoraphobia than in uncomplicated panic disorder and nonpanic anxiety disorder.

II. Determine whether the prevalence of abnormalities on audiological tests of cochlear or brainstem function is elevated in panic disorder without agoraphobia or nonpanic anxiety disorder.

III. Determine whether symptom patterns can be identified that are indicative of vestibular abnormalities in panic disorder.

IV. Determine whether vestibular dysfunction can be induced by psychosomatic mechanisms.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are stratified by otoneurological function (panic disorder without agoraphobia, panic disorder with agoraphobia, anxiety disorder without panic or agoraphobia-like avoidance, and normal controls).

Patients undergo a psychiatric interview and a structured interview focused on anxiety disorders. Physical evaluation is completed.

A vestibular evaluation consisting of posturography, rotational testing, and ocular motor screening battery, and positional and caloric testing is completed on all patients. Patients then complete an audiological test battery consisting of basic audiological analysis, speech recognition scores, immittance testing, brainstem evoked response, and determination of binaural masking level differences.

Control patients also complete a hyperventilation-rotational test.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnostically proven panic disorders with or without moderate or severe agoraphobia and anxiety disorders without panic or agoraphobia Panic disorder may be accompanied by a secondary Axis 1 diagnosis of another disorder, such as depression, generalized anxiety disorder, or dependent, histrionic, or compulsive personality disorder --Prior/Concurrent Therapy-- Surgery: No prior ear surgery Other: No concurrent medication for medical or psychiatric conditions At least 2 weeks since prior medication No ototoxic drug intake --Patient Characteristics-- No medical disorders At least 2 weeks since prior upper respiratory tract infection and recovered No history of migraine No head trauma No scoliosis No alcoholism No drug abuse No family history of schizophrenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Rolf G. Jacob, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States